CLINICAL TRIAL: NCT06055660
Title: Expression and Distribution of Membrane-Organizing Extension Spike Protein (Moesin/ MSN) is Associated With Epithelial-Mesenchymal Transition in Clear Cell Renal Cell Carcinoma.
Brief Title: Moesin Expression in Clear Cell Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, Maisa H Mohammed, MD, Sohag University
Other Study IDs: Soh-Med-23-09-5PD
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Moesin; Epithelial-Mesenchymal Transition
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Immunohistochemical detection of Moesin in Clear cell Renal Cell Carcinoma — Formalin-fixed paraffin-embedded renal cell carcinoma tissue blocks will be sectioned and immunohistochemically stained by anti moesin antibody.

SUMMARY:
Renal cell carcinoma (RCC) is the most frequently occurring primary renal neoplasm. There are several histological variants of RCC that are associated with variable prognostic outcomes. Epithelial-mesenchymal transition (EMT) is a phenomenon in which the epithelial cells acquire some mesenchymal criteria as enhanced invasive potential. There are several cell surface molecules that are implicated in EMT. Moesin is one of these molecules that is involved in EMT, which is associated with enhanced invasive potential and poor prognosis. Targeting Moesin by novel therapeutic agents may prevent EMT and improve prognosis of patients with RCC.

ELIGIBILITY:
Inclusion Criteria:

1. All cases of ccRCC.
2. Tissue blocks with material adequate for immunohistochemical evaluation.
3. All cases with accessible clinical data.

Exclusion Criteria:

1. Cases of renal neoplasms other than ccRCC.
2. Patients who received preoperative chemotherapy or radiotherapy.
3. Patients with ccRCC who were diagnosed by tru-cut biopsies only and didn't undergo radical operations.
4. Cases with insufficient/destructed material.
5. Patients with inadequate clinical data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The present work will be performed on archived formalin-fixed, paraffin-embedded renal cell carcinoma tissue blocks that were belonged to 55 patients who were admitted to Sohag University Hospital because of loin/ back pain, from January 1st,2017 to December 31st, 2021. Radiological evaluation revealed renal neoplasms and patients underwent radical nephrectomies.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of Moesin in renal cell carcinoma | 6 months
  different levels of moesin expression will be correlated with some tumor characteristics as patients' ages, sexes, tumor site, tumor grades, stages and nodal statuses.

IPD SHARING:
Plan to Share IPD: Undecided